CLINICAL TRIAL: NCT00130767
Title: Kinetics of the Finasteride Prostate Induced Apoptosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.316
Record Dates: First submitted 2005-08-12; First posted 2005-08-16 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostate; apoptosis; finasteride kinetics
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Finasteride

INTERVENTIONS:
Drug: finasteride

SUMMARY:
The aim of this study is to evaluate the mechanisms involved in the apoptosis induced by a treatment of finasteride on benign prostate hyperplasia (BPH). Five sets of patients who need a surgical procedure because of low tract urinary symptoms are randomly attributed to one of five sets of treatment: 0, 7, 14, 21 or 28 days of finasteride treatment before the day of the procedure. Prostate histological fragments are conditioned for molecular and histologic studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low tract urinary symptoms needing a surgical procedure
* No previous treatment with finasteride
* No androgen deficiency; no prostate cancer suspected.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-12

PRIMARY OUTCOMES:
Date of the maximum apoptosis in the prostate tissues treated by finasteride

SECONDARY OUTCOMES:
Molecular mechanisms involved in BPH finasteride induced apoptosis
Decrease in the frequency of the hemorrhagic incidents after the surgical procedure in patients with a treatment using finasteride

CONTACTS AND LOCATIONS:
Overall Officials: Alain RUFFION, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre hospitalier Lyon Sud, Pierre-Bénite, France